CLINICAL TRIAL: NCT03708133
Title: Open-label, Randomized, Single-dose, Cross-over Study to Assess Bioequivalence Between a Single 120 mg Nifurtimox Tablet and a Newly Developed 120 mg Nifurtimox Tablet, Administered Orally Under Fed Conditions to Adult Male and Female Patients With Chronic Chagas' Disease
Brief Title: Study to Assess Bioequivalence of a New Nifurtimox Oral Tablet Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19500
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Bioequivalence
Keywords: New formulation
MeSH Terms: interventions — Nifurtimox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Treatment + Reference Treatment (Experimental): Male and female subjects with Chagas' disease will be give treatment follow below Crossover Sequence:
  1. Test treatment
  2. Reference treatment
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502)_Test; Drug: Nifurtimox (Lampit, BAYA2502)_Reference
- Reference Treatment + Test Treatment (Experimental): Male and female subjects with Chagas' disease will be give treatment follow below Crossover Sequence:
  1. Reference treatment
  2. Test treatment
  Interventions: Drug: Nifurtimox (Lampit, BAYA2502)_Test; Drug: Nifurtimox (Lampit, BAYA2502)_Reference

INTERVENTIONS:
Drug: Nifurtimox (Lampit, BAYA2502)_Test — Orally intake of 1 *120mg new formulation tablet as test treatment
Drug: Nifurtimox (Lampit, BAYA2502)_Reference — Orally intake of 1 *120mg current clinical formulation tablet as reference treatment

SUMMARY:
The primary objective of the current study is to investigate the bioequivalence of a newly developed 120 mg nifurtimox tablet formulation (Test treatment) compared with the 120 mg nifurtimox tablet currently used in the Bayer pediatric clinical development program (Reference treatment). The new tablet formulation assessed in this study is intended to replace the 120 mg nifurtimox tablet formulation currently used in clinical practice. It is an immediate-release tablet with an altered composition compared to the reference formulation. The new tablet overcomes pharmaceutical quality issues seen for the current formulation, e.g. sensitivity to humidity. Due to safety reasons, the study drug will be administered under fed conditions to adult male and female patients suffering from Chagas' disease and not healthy subjects (see also Benefit-risk assessment below).

In addition, the PK, safety, and tolerability of nifurtimox will be assessed as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

- Male/female patient diagnosed with chronic Chagas' disease: Previous diagnosis of acute or chronic Chagas' disease by a health clinic prior to screening for the study. The diagnosis of chronic Chagas' disease may be made by clinical findings, supported by antibody titers if available. If there is a known history of acute disease, it is preferable to have documentation of parasites on the blood smear, if available.

* Women and men of reproductive potential must agree to use adequate contraception when sexually active. This applies for the time period between signing of the informed consent form and 12 weeks after the last administration of study drug. The definition of adequate contraception will be based on the judgment of the investigator and on local requirements. Acceptable methods of contraception include, but are not limited to: (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception. Subjects must agree to utilize two reliable and acceptable methods of contraception simultaneously.
* Women of childbearing potential with confirmed last menstrual period by anamnesis and negative serum pregnancy test (beta-human chorionic gonadotropin [βhCG]) at screening and negative urine pregnancy test (βhCG) at pre-dose of each treatment.
* Women of non-childbearing potential, such as surgically sterile women with either written documentation of surgical sterility or negative serum pregnancy test (βhCG) at screening and negative urine pregnancy test (βhCG) at pre-dose of each treatment.
* Male subjects who agree not to act as sperm donors for 12 weeks after last administration of study drug.
* Age: 18 to 45 years (inclusive) at screening.
* Body mass index (BMI): ≥18 and <29.9 kg/m².
* At least 3 months since delivery or abortion, or 3 months since cessation of lactation before screening.
* Ability to understand and follow study-related instructions.

Exclusion Criteria

* Acute Chagas' disease. (During the acute phase, the parasite on a blood smear may be seen under a microscope. Different antibodies are present, depending on the course of the disease).
* Known hypersensitivity to the study drug (active substance or excipients of the preparations)
* Suspected or known porphyria.
* Clinically significant allergies (e.g. allergies affecting the lower respiratory tract such as allergic asthma or allergies requiring therapy with systemic corticosteroids) within 1 year.
* Clinically significant non-allergic drug reactions, or multiple severe drug allergies (e.g. adverse reactions in the form of bronchospasm, asthma, rhinitis or urticaria after taking non-steroidal anti-inflammatory drugs).
* Unstable or uncontrolled medical condition such as hypertension or diabetes, decompensated heart failure, GI conditions that would interfere with the absorption of the study drug (e.g. GI ulceration, peptic ulceration, GI bleeding, gastroesophageal reflux, or other GI disease affecting gastroesophageal junction), conditions that could potentially have an impact on drug metabolism or elimination (renal, hepatic such as known hepatic or biliary abnormalities), or any clinically relevant active infections in the opinion of the investigator within 4 weeks before the screening visit, e.g. clinically relevant history or presence of significant respiratory (e.g. interstitial lung disease), hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, metabolic (e.g. diabetes), and dermatological or connective tissue disease.
* Incompletely cured pre-existing diseases (except chronic Chagas' disease without active GI condition) for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the study drugs will not be normal.
* Febrile illness within 1 week before the first study drug administration.
* Systolic blood pressure <100 or >140 mmHg (after resting in supine position for a minimum of 15 minutes).
* Diastolic blood pressure <50 or >90 mmHg (after resting in supine position for a minimum of 15 minutes).
* Heart rate <45
* Positive pregnancy test.
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV), or human immunodeficiency virus antibodies (anti-HIV 1+2).
* Positive urine drug screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
AUC of nifurtimox in plasma | Pre-dose (up to 30 minutes before study drug administration), and at 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 hours post-dose
  AUC:area under the concentration versus time curve from zero to infinity after single (first) dose
AUC(0-tlast) of nifurtimox in plasma | Pre-dose (up to 30 minutes before study drug administration), and at 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 hours post-dose
  AUC(0-tlast): AUC from time 0 to the last data point > LLOQ(lower limit of quantitation)
Cmax of nifurtimox in plasma | Pre-dose (up to 30 minutes before study drug administration), and at 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 hours post-dose
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration

SECONDARY OUTCOMES:
tmax of nifurtimox in plasma | Pre-dose (up to 30 minutes before study drug administration), and at 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 hours post-dose
  tmax: time to reach Cmax
t1/2 of nifurtimox in plasma | Pre-dose (up to 30 minutes before study drug administration), and at 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 hours post-dose
  t1/2: Half-life associated with terminal slope
AUCnorm of nifurtimox in plasma | Pre-dose (up to 30 minutes before study drug administration), and at 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 hours post-dose
  AUCnorm: AUC divided by dose per body weight
Cmax,norm of nifurtimox in plasma | Pre-dose (up to 30 minutes before study drug administration), and at 15 minutes, 30 minutes, 45 minutes, and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 15 hours post-dose
  Cmax,norm: Cmax divided by dose per body weight
Number of participants with treatment emergent adverse events | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- FP Clinical Pharma, Buenos Aires, Ciudad Auton. de Buenos Aires, Argentina